CLINICAL TRIAL: NCT07040436
Title: REVERT Study: A Phase 1b/2a Study to Assess the Safety and Efficacy of OPM-101 Combined With Anti-PD-1 in Patients With Advanced Melanoma Showing Resistance to Anti-PD-1
Brief Title: Assessment of Safety and Efficacy of OPM-101 Combined With Anti-PD-1 in Patients With Advanced Melanoma Showing Resistance to Anti-PD-1
Acronym: REVERT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncodesign Precision Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPM101-P2-01
Record Dates: First submitted 2025-06-13; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Advanced Melanoma
Keywords: OPM-101; Melanoma; resistance; Anti-PD1; RIPK2; advanced; immuno-oncology; anti-PD1 refractory; pembrolizumab
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Open label phase 1b/2a study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPM-101 (in combination with pembrolizumab) (Experimental): OPM-101 will be administered as hard gelatin capsules twice a day for 24 weeks. In the Phase 1b, 2 doses of OPM-101 will be considered: 75 mg bid and 150 mg bid. At the end of this Phase 1b, a recommended dose for Phase 2a will be determined. During the Phase 2a, the recommended dose of OPM-101 will be administered bid over 24 weeks.
  OPM-101 will be administered in combination with authorized regimen of Pembrolizumab.
  Interventions: Drug: OPM-101

INTERVENTIONS:
Drug: OPM-101 — OPM-101 will be administered in combination with an authorized regimen of Pembrolizumab.
  Pembrolizumab will be administered by IV infusion either at a dose of 200 mg every 3 weeks or at a dose of 400 mg every 6 weeks, as per Principal Investigator's decision.

SUMMARY:
This is a phase 1b/2a study including a dose escalation part (Phase 1b) and an extension part (Phase 2a).

Both parts will be open-label, multicenter study of OPM-101 combined with the anti-PD-1 pembrolizumab as per standard of care in patients with MM who have been receiving an anti-PD-1-based treatment and have shown resistance to it, as defined by the Society for Immunotherapy of Cancer (SITC) criteria (Kluger, 2020). The objective of the study is to assess whether the addition of OPM-101 will resensitisze the tumour to the anti-PD-1-based treatment.

Potential patients will be screened for this study during the period between initial evidence of disease progression on anti-PD-1 treatment and the required radiographic confirmation of disease progression. The intent is to initiate treatment with OPM-101 once the suspicion of disease progression on anti-PD-1-based therapy is confirmed, and the patient has signed the study Information and Consent Form. No anti-PD-1-based treatment should be administered within 4 weeks prior to study treatment initiation.

In the dose escalation part (Phase 1b) of the study, two different doses of OPM-101 will be evaluated (75 mg bid and 150 mg bid) in combination with pembrolizumab. Patients will receive the dose and regimen of pembrolizumab, as per the authorised product SmPC, in sequential cohorts using a 3 + 3 design, escalating if 0 of 3 (or 1 of 6) patients experience a dose-limiting toxicity (DLT) during the first 6 weeks of treatment and not escalating if 2 of 6 patients experience a DLT.

The RP2D of OPM-101 for the second part of the study (Phase 2a) in combination with pembrolizumab will be based on the rate of DLTs, incidence and severity of Treatment-Related AEs (AEs) and SAEs, and frequency of dose holds, reductions and discontinuations.

A Data and Safety Monitoring Board (DSMB) will assess the safety criteria and make recommendations about dose escalation/de-escalation during the Phase 1b part, and on the RP2D to be used for further patients in the Phase 2a. The selection of the dose level for the Phase 2a will be based on safety and on preliminary PK/PD or even trends of efficacy. The DSMB will also review periodically the data during the Phase 2a and make recommendations about the continuation of the study.

The cohort expansion part (Phase 2a) of the study will be conducted once the Phase 1b is completed and a safe and tolerated dose (potentially 150 mg bid) has been determined. Patients will receive daily oral treatment with OPM-101, while taking pembrolizumab for at least 12 weeks, i.e., at the time of the radiographic assessment of the disease for the primary endpoint evaluation. Patients who show a treatment response with Disease Control (CR, PR or SD) at 12 weeks will continue treatment with [OPM-101 + pembrolizumab] up to 24 weeks, when the second radiographic disease assessment is performed.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent provided prior to any study-related procedure.
2. Histologically confirmed, unresectable or metastatic stage III or IV melanoma.
3. At least one measurable lesion per RECIST v.1.1 criteria.
4. Patients with a documented and confirmed Progressive Disease with an anti-PD-1-based treatment given alone or in combination (except combination with an anti-LAG-3 drug). Progressive disease will be determined by the PI based on the SITC v3.0 guidelines.

   Note: Patients who have been treated with a combination of nivolumab and ipilimumab will also be considered for study inclusion.
5. Patients with no anti-PD-1-based treatment administration within 4 weeks (or 6 weeks for a treatment with pembrolizumab administered with a 400 mg q6w scheme) prior to study treatment initiation.
6. Patients accepting to undergo a fresh biopsy at baseline and after 12 weeks of treatment (for Phase 1b only).

   * In case a fresh baseline biopsy collection would represent a medical risk for the patient, an archival biopsy could be used, after discussion with the Medical Monitor and the Principal Investigator (PI)
   * If archival sample is unavailable, and the patient cannot provide a fresh tumour biopsy at baseline due to medical risk or inaccessibility, the patient may still be enrolled if agreed upon between the Investigator and the Sponsor.
7. Male or female patients ≥18 years.
8. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
9. Estimated life expectancy ≥3 months.
10. Adequate hematologic parameters and organ function defined by:

    * white blood cell count ≥3,000/µL
    * absolute neutrophil count ≥1,500/µL without support of filgrastim
    * platelet count ≥75,000/µL
    * haemoglobin (Hgb) ≥9 g/dL (criterion must be met without erythropoietin dependency and without packed red blood cell transfusion within last 2 weeks)
    * calculated creatinine clearance ≥50 mL/min (Cockroft Gault formula)
    * serum total bilirubin ≤1.5 x ULN (or ≤3.0 x ULN if documented Gilbert syndrome) analysed using vanadate method.
    * AST and ALT ≤2.5 x ULN (or ≤5.0 x ULN if liver metastases)
    * International normalized ratio (INR) ≤1.5 x ULN unless patient is receiving anticoagulant therapy if partial thromboplastin or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
    * Urinalysis negative for haematuria
11. Females of childbearing potential must have confirmed negative pregnancy test prior to OPM-101 administration (daily oral dosing) and willing to use effective contraception during OPM-101 treatment and for at least 3 months after the last dose of OPM-101. Females considered of non-childbearing potential are post-menopausal women and women having undergone hysterectomy.
12. Females with childbearing potential must not be breast feeding.
13. Males must agree to use effective barrier contraception during OPM-101 treatment and for 90 days (a spermatogenesis cycle) after the last dose of OPM-101.

Exclusion criteria

1. Diagnosis of primary uveal and/or ocular melanoma, as well as mucosal melanoma
2. Active leptomeningeal disease or uncontrolled brain metastasis. Patients with equivocal findings or with confirmed brain metastases are eligible for enrolment provided they are asymptomatic without the need for corticosteroid treatment for at least 4 weeks prior to the first dose of study drug(s).
3. Patients who have received any line of therapy with a BRAF inhibitor or MEK inhibitor in the advanced disease setting.
4. Treatment with any of the following anti-cancer therapies prior to the first dose of study treatment within the stated timeframes:

   * 4 weeks for any anti-PD-1-based therapy (except for previous treatments with pembrolizumab administered with a 400 mg q6w scheme for which the duration should be 6 weeks)
   * 4 weeks for radiation therapy
   * 2 weeks for limited field radiation for palliation
   * 4 weeks or 5 half-lives (whichever is longer) for continuous or intermittent small molecule therapeutics or any other investigational agent, receiving study therapy or has participated in a study of an investigational agent and received study therapy, or used an investigational device. The participation in the follow-up Phase (i.e., receiving no study treatment) of a prior study is allowed.
   * 6 weeks for cytotoxic agents with major delayed toxicities, such as nitrosoureas and mitomycin C
5. History of severe or life-threatening immune-related (IR) AEs during a previous treatment with anti-PD-1

   * IR-myocarditis
   * Grade ≥3, IR- interstitial lung disease IR-renal toxicity.
   * Grade 4 for IR-maculopapular rash, IR-diarrhoea and enterocolitis, IR-rheumatological toxicity, IR-neuro(muscular) toxicity, IR-hepatotoxicity
6. Unrecovered CTCAE at time of screening

   * Any patient unrecovered to a CTCAE grade ≤2 for patients who has been pre-treated with anti-PD-1 monotherapy
   * Any patient unrecovered to a CTCAE grade ≤ 1 for patients who has been pre-treated with the combination of nivolumab plus ipilimumab
7. Any of the following cardiovascular criteria:

   * Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤28 days before the first dose of study drug(s)
   * Symptomatic pulmonary embolism ≤28 days before the first dose of study drug(s)
   * Any history of acute myocardial infarction ≤6 months before the first dose of study drug(s)
   * Any history of heart failure meeting New York Heart Association Classification (NYHA) class III or IV ≤6 months before the first dose of study drug(s)
   * Any event of ventricular arrhythmia ≥Grade 2 in severity ≤6 months before the first dose of study drug(s)
   * Any history of cerebrovascular accident ≤6 months before the first dose of study drug(s)
   * Uncontrolled hypertension: systolic pressure ≥160 mmHg or diastolic pressure ≥100 mmHg despite anti-hypertension medications ≤28 days before the first dose of study drug(s)
   * Any episode of syncope or seizure ≤28 days before the first dose of study drug(s)
8. Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤4 weeks before administration of study drug.

   Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:
   * Adrenal replacement steroid (dose ≤10 mg daily of prednisone or equivalent)
   * Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
   * Short course (≤7 days) of corticosteroid prescribed prophylactically, e.g., for contrast dye allergy, or for the treatment of a non-autoimmune condition, e.g., delayed-type hypersensitivity reaction caused by contact allergen
9. Active infection requiring systemic therapy
10. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
11. Active autoimmune diseases or history of autoimmune diseases that may relapse. Patients with the following diseases are not excluded and may proceed to further screening:

    * Controlled type 1 diabetes
    * Hypothyroidism provided it is managed with hormone replacement therapy only
    * Controlled celiac disease
    * Skin diseases not requiring systemic treatment, e.g., vitiligo, psoriasis, alopecia
    * Any other disease that is not expected to recur in the absence of external triggering factors
12. Known history of Human Immunodeficiency Virus (HIV, HIV 1/2 antibodies), known active Hepatitis B, i.e., HBsAg positive or detectable HBV DNA, known active Hepatitis C, i.e., detectable HCV RNA (qualitative).
13. Hypersensitivity to any excipients in OPM-101 formulation, i.e., lactose, cellulose, polyvinylpyrrolidone, magnesium stearate.
14. Hypersensitivity to any excipients in the pembrolizumab formulation (L-histidine, L-histidine hydrochloride monohydrate, sucrose, polysorbate 80)
15. Patients who received live vaccine within 30 days of planned start of the study therapy.
16. History or current evidence of any condition, therapy, laboratory abnormality or psychiatric or substance abuse disorder that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Patients who received homeopathy within 14 days of planned start of the study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the recommended dose | 6 weeks
  In the phase 1b: the recommended dose for phase 2a will be based on the independent assessement of safety of OPM-101 by the DSMB
Determination of the Disease Control Rate (DCR) | 12 weeks
  In phase 2a, Disease Control Rate defined as CR, PR or SD as per RECIST v.1.1 criteria

SECONDARY OUTCOMES:
Determination of the Disease Control Rate | 12 weeks
  In Phase 1b: Disease Control Rate (DCR= CR+PR+SD) per RECIST v.1.1 criteria.
Determination of the Disease Control Rate | 24 weeks
  In Phase 1b and Phase 2a: Disease Control Rate (DCR= CR+PR+SD) per RECIST v.1.1 criteria.
Determination of the objective response rate (ORR) | Week 12 and Week 24
  In the phase 1b and Phase 2a, the objective response rate (ORR = CR + PR) will be evaluated using RECIST v1.1 criteria
Determination of the frequency of dose reduction, and discontinuations | 24 weeks
  In Phase 1b and Phase 2a
Safety assessments | 24 weeks
  Phase 2a: determine the incidence and severity of adverse events (AEs) and serious adverse events (SAEs

OTHER OUTCOMES:
Biomarker: Cytokine evaluation | 24 weeks
  In Phase 1b and Phase 2a, measurement of circulating cytokines. A panel of cytokines known to be regulated by immune responses and by the RIPK2 pathway will be assessed
Biomarker: Chemokine evaluation | 24 weeks
  In Phase 1b and Phase 2a, measurement of circulating chemokines. A panel of chemokines known to be regulated by immune responses and by the RIPK2 pathway will be assessed.
Pharmacokinetics parameters (Cmax) | Day 1
  In phase 1b only, determination of the Maximal concentration (Cmax) after the first OPM-101 treatment intake
Pharmacokinetics parameters (Cmin) | Day 2, Week 6 and Week 12
  In phase 1b only, measurement of the residual conentration (Cmin) 24h after the first OPM-101 treatment intake (i.e., on Day 2) and at Week 6 and Week 12
Pharmacokinetics parameters (Tmax) | Day 1
  In phase 1b only, determination of the time to reach the Maximal concentration (Tmax) after the first OPM-101 treatment intake
Pharmacokinetics parameters (AUC0-24) | Day 1
  In phase 1b only, determination of the systemic exposure (Area Under the Curve - AUC 0-24) to OPM-101 calculated over 24h after the first OPM-101 treatment intake
Pharmacodynamics (target engagement) | Day 1
  In phase 1b only, measurement of target engagement measured by the stimulated TNFalpha production at pre-dose (T0) and 1, 2-, 4-, 8- and 24-hours after the first OPM-101 dosing on Day 1.